CLINICAL TRIAL: NCT01284023
Title: Use of Near Infrared Spectroscopy to Detect Muscle Perfusion in the Lower Extremity of Uninjured Subjects
Status: Completed | Type: Observational
Sponsor: J&M Shuler (Industry)
Collaborators: Nonin Medical, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: NIRS-02
Record Dates: First submitted 2011-01-25; First posted 2011-01-26 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Acute Compartment Syndrome
Keywords: near infrared spectroscopy; acute compartment syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Controls: Uninjured volunteers
  Interventions: Other: Shaving

INTERVENTIONS:
Other: Shaving — Male patients will have the leg hair under each sensor site shaved, using an electric razor, and near infrared spectroscopy monitored for an additional 15 minutes

SUMMARY:
Acute compartment syndrome (ACS) is a complication of lower leg trauma that occurs when the pressure inside the leg due to swelling exceeds the body's ability to provide blood to the muscle of the leg. This condition cuts off blood flow to the leg. Left untreated, the condition can result in devastating consequences including complete loss of function of the lower extremity or amputation. Near-infrared spectroscopy (NIRS)-based tissue perfusion monitors are a non-invasive means of continuously monitoring the amount of oxygen in the tissues of an injured extremity. The device utilizes harmless red light to detect the proportion of hemoglobin saturated with oxygen up to 3 cm below the skin surface. The purpose of this study will be to launch the first stages of validation of this device as a diagnostic tool for compartment syndrome, by observing this device in uninjured subjects.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old

Exclusion Criteria:

* any current traumatic lower or upper extremity injury
* unwilling or unable to provide written informed consent
* history of any anatomy-altering injury or procedure to the upper or lower extremity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Uninjured volunteers will be recruited from a pool of uninjured individuals at the principle investigator's practice. Participation will be completely volutnary
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Near infrared spectroscopy | 1 hour
  Uninjured subjects will lay supine and be monitored for two one hour periods, on separate days.

SECONDARY OUTCOMES:
Skin pigmentation | prior to monitoring
  due to absorption of hemoglobin and melanin at near infrared wavelengths, skin pigmentation may affect near infrared spectroscopy values. Skin pigmentation values will be recorded on each study participant using the DSM-II (CyberDerm, Broomall, PA) and the IMS SmartProbe (IMS, Portland, ME).
fat depth | prior to monitoring
  because the near infrared spectroscopy device measures tissue oxygenation 2-3 cm below the skin, the device may obtain an altered reading or be unable to obtain a reading on subjects with excessive subcutaneous fat. Data on fat depth will be collected on control subjects using the BX2000 (IntelaMetrix, Livermore, CA)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Shuler, MD, Principal Investigator — Athens Orthopedic Clinic, PA
Locations (1):
- Athens Orthopedic Clinic, PA, Athens, Georgia, United States